CLINICAL TRIAL: NCT01236768
Title: An Open-Label, Randomized, Phase 3 Study of the Contraceptive Efficacy and Safety of Agile Transdermal Contraceptive Delivery System in Comparison to an Oral Contraceptive (OC) Containing 150 mcg LNG and 30 mcg EE
Brief Title: Transdermal Contraceptive Delivery System (TCDS), Also Known as AG200-15 Patch Arm
Acronym: ATI-CL13
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Agile Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ATI-CL13
Record Dates: First submitted 2010-11-05; First posted 2010-11-09 (Estimated); Results first posted 2017-09-15 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-08

CONDITIONS: Contraception
Keywords: Contraceptive
MeSH Terms: interventions — Ethinyl Estradiol-Norgestrel Combination; Contraceptives, Oral, Hormonal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AG200-15 (Experimental): Thin transdermal contraceptive delivery system (TCDS) that gives systemic exposure of levonorgestrel (LNG) and ethinyl estradiol (EE)
  Interventions: Drug: AG200-15
- Levora (Active Comparator): oral contraceptive containing 150mcg of LNG and 30mcg of EE
  Interventions: Drug: Levora

INTERVENTIONS:
Drug: AG200-15 — Contraception; AG200-15 is applied and replaced every 7 days for 3 weeks, followed by a 1-week "patch free" period.
  Other Names: Transdermal contraceptive delivery system (TCDS)
  Arms: AG200-15
Drug: Levora — One tablet of Levora will be taken each day for a 28 day cycle.
  Other Names: Hormonal oral contraceptive
  Arms: Levora

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of a low dose transdermal contraceptive delivery system containing ethinyl estradiol and levonorgestrel.

DETAILED DESCRIPTION:
Comparative evaluation of AG200-15 versus OC with regard to safety, contraceptive efficacy, hormone related adverse events, lipid profile, cycle control (bleeding pattern), subject compliance and serum concentrations of EE and LNG. To evaluate TCDS wearability (including adhesion).

ELIGIBILITY:
Inclusion Criteria:

* sexually active women requesting contraception
* Regular menses every 24 - 35 days
* In good general health, confirmed by medical history, physical (including gynecologic examination adn screening laboratory values

Exclusion Criteria:

* Known or suspected pregnancy
* Lactating women
* Significant skin reaction to transdermal preparations or sensitivity to surgical / medical tape
* Any disease that may worsen under hormonal treatment (cardiovascular, liver, metabolic)
* Use of other contraceptive methods than study medication

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 407 (Actual)
Dates: Start 2010-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie Foegh, MD, Study Director — Agile Therapeutics
Locations (19):
- United States (19):
  - Mobile, Alabama
  - Green Valley, Arizona
  - Tucson, Arizona
  - Los Angeles, California
  - West Hills, California
  - Boynton Beach, Florida
  - South Miami, Florida
  - St. Petersburg, Florida
  - Newburgh, Indiana
  - Louisville, Kentucky
  - Las Vegas, Nevada
  - Kernersville, North Carolina
  - Englewood, Ohio
  - Tulsa, Oklahoma
  - Mt. Pleasant, South Carolina
  - Corpus Christi, Texas
  - Sugar Land, Texas
  - Newport News, Virginia
  - Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- AG200-15: Transdermal contraceptive delivery system (TCDS)
- Levora: hormonal oral contraceptive
Period: Overall Study
Arm/Group | AG200-15 | Levora
Started | 201 | 206
Completed | 112 | 145
Not Completed | 89 | 61

BASELINE CHARACTERISTICS:
Population: Safety Population (number of subjects that received drug)
Groups:
- Total: Total of all reporting groups
Arm/Group | AG200-15 | Levora | Total
Number analyzed (Participants) | 177 | 188 | 365
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 177 | 188 | 365
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 177 | 188 | 365
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 177 | 188 | 365

OUTCOME MEASURES:

1. Primary Outcome: Pregnancy Reported as Pearl Index
Description: Pearl Index is the number of on-therapy pregnancies times 1300 divided by the number of 28-day on-therapy cycles and is an estimate of the number of pregnancies per 100 woman-years of product use.
Time Frame: 6 months
Population: Intent-to-treat population ages 18-35.
Measure: Number (95% Confidence Interval); unit: Pearl Index
Arm/Group | AG200-15 | Levora
Number analyzed (Participants) | 147 | 163
Pearl Index | 8.19 [0.19 to 16.19] | 6.80 [0.15 to 13.44]

2. Secondary Outcome: Safety
Description: Adverse events
Time Frame: 6 months
Population: Any subject who applied a patch.
Measure: Number; unit: Events
Arm/Group | AG200-15 | Levora
Number analyzed (Participants) | 177 | 188
Events | 85 | 88

3. Other Pre Specified Outcome: Cycle Control
Description: The percentage of cycles with breakthrough bleeding or spotting episodes during all cycles. Numerator is total number of cycles with event, denominator is total number of cycles.
Time Frame: 6 months
Population: Subjects with relevant breakthrough bleeding (BTB) and/or spotting (BTS), and drug information for a cycle.
Measure: Number; unit: percent cycles with BTB or BTS
Arm/Group | AG200-15 | Levora
Number analyzed (Participants) | 162 | 182
percent cycles with BTB or BTS | 24.5 | 21
Statistical Analysis 1: Comparison: AG200-15 vs Levora; Comparative evaluation of AG200-15 and Levora; Test type: Equivalence — Comparative analysis of AG200-15 and Levora for breakthrough bleeding and/or spotting; p = 0.089, Chi-squared

4. Other Pre Specified Outcome: Irritation and Itching at Application Site
Description: AG200-15 irritation and itching scores are defined as follows:
  0=none
  1. mild
  2. moderate
  3. severe
Time Frame: 6 months
Population: Subject self-reported worse irritation score in a cycle.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | AG200-15
Number analyzed (Participants) | 170
Score
  Irritation Score (cycles 1-6 combined) | 1.15 (0.914)
  Itching Score (cycles 1-6 combined) | 1.31 (0.851)

5. Other Pre Specified Outcome: Pharmacokinetics of Levonorgestrel (LNG) and Ethinyl Estradiol (EE)
Description: Measurement of plasma levels of levonorgestrel and ethinyl estradiol.
Time Frame: 3 months and 6 months
Population: Number of subjects with available LNG data for cycle 3 or cycle 6
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | AG200-15 | Levora
Number analyzed (Participants) | 111 | 140
pg/mL
  LNG cycle 3 | 2244 [1887 to 2600] | 3474 [3044 to 3904]
  LNG cycle 6 | 1743 [1478 to 2007] | 3682 [3136 to 4228]
  EE cycle 3 | 44.5 [38.7 to 50.3] | 50.6 [43.0 to 58.3]
  EE cycle 6 | 34.7 [30.1 to 39.4] | 54.7 [44.8 to 64.5]

6. Other Pre Specified Outcome: Adhesion at Application Site
Description: Measurement of adhesion of application site is defined as follows:
  0: >=90% adhered (no lifting)
  1. >=75% adhered but <90% (some edges showing lifting)
  2. >=50% adhered but <75% (half of the patch lifts off)
  3. <50% (> half of patch lifts off, but not detached)
  4. patch completely detached
Time Frame: 6 months
Population: Subjects that have documented adhesion scores.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | AG200-15
Number analyzed (Participants) | 159
Score | 0.46 (1.118)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | AG200-15 | Levora
All-Cause Mortality (participants affected / at risk) | 0/177 | 0/188
Serious Adverse Events (participants affected / at risk) | 0/177 | 2/188
Other Adverse Events (participants affected / at risk) | 42/177 | 45/188
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AG200-15 (N=177) | Levora (N=188)
Murine Typhus (Infections and infestations) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AG200-15 (N=177) | Levora (N=188)
Nausea (Gastrointestinal disorders) | 5 (5) | 11 (11)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 8 (8)
Sinusitis (Infections and infestations) | 7 (7) | 5 (5)
Cervical dysplasia (Reproductive system and breast disorders) | 10 (10) | 11 (11)
Nasopharyngitis (Infections and infestations) | 9 (9) | 8 (8)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Review and approval by Agile Therapeutics, Inc. of any publication, including oral presentations and abstracts, utilizing data or any information from the ATI-CL13 study is required prior to publication submission.